CLINICAL TRIAL: NCT02150759
Title: Comparison Study of Analgesic Effects for Dexmedetomidine-fentanyl vs Dexmedetomidine-ketamine in Femur Proximal Fracture Patients
Brief Title: Dexmedetomidine-ketamine in Femur Proximal Fracture Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Ki Hwa Lee, Assistant professor, Inje University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2014-027
Record Dates: First submitted 2014-05-23; First posted 2014-05-30 (Estimated); Results first posted 2019-04-29 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Pain
Keywords: Dexmedetomidine; Ketamine; Pain
MeSH Terms: conditions — Pain | interventions — Dexmedetomidine; Fentanyl; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexmedetomidine-ketamine (Experimental): Dexmedetomidine-ketamine group
  Interventions: Drug: Dexmedetomidine; Drug: Ketamine
- Dexmedetomidine-fentanyl (Active Comparator): Dexmedetomidine-fentanyl group
  Interventions: Drug: Dexmedetomidine; Drug: Fentanyl

INTERVENTIONS:
Drug: Dexmedetomidine — dexmedetomidine infusion during spinal anesthesia
  Other Names: Precedex
Drug: Fentanyl — add dexmedetomidine during position change
  Other Names: fentanyl citrate
  Arms: Dexmedetomidine-fentanyl
Drug: Ketamine — add dexmedetomidine during position change
  Other Names: ketamine HCl
  Arms: Dexmedetomidine-ketamine

SUMMARY:
* Comparison study of analgesic effects for dexmedetomidine-fentanyl vs dexmedetomidine-ketamine
* lateral position for spinal anesthesia in femur proximal fracture patients

DETAILED DESCRIPTION:
* Dexmedetomidine (1mcg/kg)- fentanyl (1mcg/kg) vs dexmedetomidine (1mcg/kg) - ketamine (1mg/kg) 10 minutes loading.
* After 10 minutes of drug infusion, patients are prepared for spinal anesthesia.
* pain scale and quality of patient positioning are measured three times (lateral position, chest-knee position, intrathecal local anesthetics injection)
* When patients have severe pain during intraoperative period, fentanyl 50 mcg will be intravenously inject.
* Patients will be injected propofol 10mg when they have agitation signs during operation.
* vital signs, bispectral index, korean version of mini mental status examination, verbal rating scale,fentany/propofol consumption, frequency of intrathecal injection

ELIGIBILITY:
Inclusion Criteria:

* American society of anesthesiologists classification 1-3 patients
* >20 years old

Exclusion Criteria:

* patients refuse
* dementia patients, cooperation difficult patients
* anaphylaxis of dexmedetomidine, ketamine, local anesthetics
* heart problem (bradycardia, atrioventricular block)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-05; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sang Eun Lee, MD, Study Chair — Inje University
Locations (1):
- Haeundae paik hospital, inje university, Busan, South Korea

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: from May 2014 to October 2016
Period: Overall Study
Arm/Group | Dexmedetomidine-ketamine | Dexmedetomidine-fentanyl
Started | 23 | 23
Completed | 22 | 21
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Dexmedetomidine-Ketamine: Dexmedetomidine-Ketamine combination
- Dexmedetomidine-Fentanyl: Dexmedetomidine-Fentanyl combination
- Total: Total of all reporting groups
Arm/Group | Dexmedetomidine-Ketamine | Dexmedetomidine-Fentanyl | Total
Number analyzed (Participants) | 22 | 21 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.28 (6.47) | 79.57 (7.13) | 78.90 (6.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 14 | 34
  Male | 2 | 7 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 22 | 21 | 43
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 21 | 22 | 43
weight [Mean (Standard Deviation); unit: kg] | 52.22 (8.67) | 55.79 (8.15) | 53.96 (8.51)

OUTCOME MEASURES:

1. Primary Outcome: Pain Score Using Five Scales
Description: We want to compare pain score (five scales; 0=calm, 1=facial grimacing, 2=moaning, 3=screaming, 4=restlessness or agitation, unable to proceed) when patients are lateral position during spinal anesthesia.
Time Frame: average 10-20 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Dexmedetomidine-ketamine | Dexmedetomidine-fentanyl
Number analyzed (Participants) | 22 | 21
Participants
  Lateral position: 0 | 15 | 0
  Lateral position: 1 | 5 | 0
  Lateral position: 2 | 2 | 5
  Lateral position: 3 | 0 | 16
  Lateral position: 4 | 0 | 0
  Hip flexion: 0 | 17 | 1
  Hip flexion: 1 | 3 | 0
  Hip flexion: 2 | 1 | 6
  Hip flexion: 3 | 1 | 14
  Hip flexion: 4 | 0 | 0
  Spinal blodk: 0 | 17 | 11
  Spinal blodk: 1 | 2 | 8
  Spinal blodk: 2 | 3 | 2
  Spinal blodk: 3 | 0 | 0
  Spinal blodk: 4 | 0 | 0

2. Secondary Outcome: Quality of Patient Positioning
Description: We estimate quality of patient positioning (0=not satisfactory, 1=satisfactory, 2=good, 3=optimal) during spinal anesthesia between two groups.
Time Frame: average 10-20 minutes during spinal anesthesia
Measure: Count of Participants; unit: Participants
Arm/Group | Dexmedetomidine-ketamine | Dexmedetomidine-fentanyl
Number analyzed (Participants) | 22 | 21
Participants
  Lateral position: 0 | 2 | 3
  Lateral position: 1 | 3 | 15
  Lateral position: 2 | 9 | 3
  Lateral position: 3 | 8 | 0
  Hip flexion: 0 | 3 | 5
  Hip flexion: 1 | 6 | 13
  Hip flexion: 2 | 5 | 3
  Hip flexion: 3 | 8 | 0
  Spinal block: 0 | 1 | 3
  Spinal block: 1 | 7 | 13
  Spinal block: 2 | 6 | 5
  Spinal block: 3 | 8 | 0

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Dexmedetomidine-Ketamine | Dexmedetomidine-Fentanyl
All-Cause Mortality (participants affected / at risk) | 0/22 | 1/21
Serious Adverse Events (participants affected / at risk) | 0/22 | 1/21
Other Adverse Events (participants affected / at risk) | 21/22 | 20/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexmedetomidine-Ketamine (N=22) | Dexmedetomidine-Fentanyl (N=21)
postoperative cardiopulmonary resuscitation (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexmedetomidine-Ketamine (N=22) | Dexmedetomidine-Fentanyl (N=21)
Bradycardia (Cardiac disorders) | 18 (18) | 14 (14)
Hypotension (Cardiac disorders) | 21 (21) | 20 (20)
desaturation (Respiratory, thoracic and mediastinal disorders) | 18 (18) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-24): https://cdn.clinicaltrials.gov/large-docs/59/NCT02150759/Prot_SAP_000.pdf